CLINICAL TRIAL: NCT03151473
Title: Prospective Cohort Assessing The Prevalence And Progress Of Non-Alcoholic Fatty Liver Disease (NAFLD)/Non-Alcoholic Steatohepatitis (NASH) In Chinese Subjects
Brief Title: Longitudinal Observational Study Of Chinese With NAFLD/NASH
Status: Recruiting | Type: Observational
Sponsor: Humanity and Health Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: H&H_NAFLD/NASH study_1
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease (NAFLD); Non-Alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum/Plasma/Liver biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a 10-year, longitudinal, observational study of patients with NAFLD/NASH designed to specifically address important clinical questions that remain incompletely answered from registration trials. In addition to the study database, the biospecimen repository will also be included so that translational studies of genomics and biomarkers of response may be performed.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is an excess accumulation of fat in the liver cells. It is associated with obesity, high blood pressure, high cholesterol, and diabetes. Some people with NAFLD only have excess fat in the liver. However, other people may develop a worse form of NAFLD with liver injury and scarring. This form, called non-alcoholic steatohepatitis (NASH), can lead to liver failure, liver cancer, and death. Not much is known about why some people develop NASH and others do not.

This study aims to determine and elucidate, through the cooperative effort of a multidisciplinary and multicenter group of collaborators, the etiology, natural history, diagnosis, treatment, and prevention of NAFLD, and in particular its more severe form of NASH and its complications in Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 and older;
* Adults being managed or treated for NAFL or NASH;
* Be able to communicate meaningfully with the Investigator and be legally competent to provide written informed consent.

Exclusion Criteria:

* Incompetent to understand and/or sign the informed consent;
* Ethanol consumption exceeding more than 14 standard beverages per week for males and more than 7 standard beverages per week for female;
* Causes for secondary hepatic fat accumulation such as significant alcohol consumption, medications, Wilson's disease, viral infections, starvation or parenteral nutrition, among others, and conditions associated with microvesicular steatosis
* Diagnosis of liver cirrhosis and/or hepatocellular carcinoma;
* Diagnosis of chronic inflammatory disease (i.e. inflammatory bowel disease, rheumatoid arthritis, inflammatory lung disease, severe infectious diseases), other than NAFL/NASH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects (BMI ≥ 25 kg/m2) with proven NAFL/NASH either by imaging (using MRI) or histology, referred to secondary or tertiary care for liver related problems will be asked to participate in this study.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NAFL/NASH in Chinese | up to 10 years
  Determine the prevalence of NAFLD/NASH in military beneficiaries ages 18 or above. This will be determined by the % of subjects determined to have NAFLD/NASH in Chinese subjects.

SECONDARY OUTCOMES:
Live imaging analysis | up to 10 years
  Transient elastography (FibroScan) and/or MR elastography will provide a measurement of liver stiffness. The liver stiffness metrics will be tabulated for each of the three time points and assessed for change.
Exploration, identification and validation of the circulating biomarkers for prediction and diagnosis of NAFL/NASH in Chinese | up to 10 years
  Cytokeratin-18 (CK-18), fibrosis-4 (FIB-4), leptin, adiponectin, TNF-alpha, PAI-1, IL-6, MCP-1, retinoids and other potential biomarkers will be determined and analysed.
Liver histology analysis | up to 10 years
  Liver histology (derived from central reading of liver biopsy at entry, standard of care biopsy done during screening or follow-up) will be examined and scored.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanity and Health Medical Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No